CLINICAL TRIAL: NCT05409222
Title: Study of Quality of Life Post Preventive Salpingo-oophorectomy in Healthy BRCA1/2 and PALB2 Mutation Carriers
Brief Title: Study of Quality of Life Post Salpingo-oophorectomy in BRCA1/2 & PALB2 Mutation Carriers (BRCA-HRT)
Acronym: BRCA-HRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ECV-2019-103
Record Dates: First submitted 2021-03-13; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Hereditary Breast and Ovarian Cancer
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1A: preventive salpingo-oophorectomy with hormone replacement therapy: Healthy carriers who decide undergo preventive surgery and opt to have hormone replacement therapy
- Cohort 1B: preventive salpingo-oophorectomy without hormone replacement therapy: Healthy carriers who decide undergo preventive surgery and reject hormone replacement therapy
- Cohort 2: without preventive salpingo-oophorectomy: Healthy carriers who decide not to proceed to preventive surgery

SUMMARY:
1. Premenopausal BRCA1 / 2 or PALB2 gene mutation carriers who receive hormone replacement therapy (HRT) after preventive salpingo-oophorectomy (PBSO) have a better quality of sexual, psychological, cardiovascular and bone health than carriers who decline HRT.
2. Premenopausal mutation carriers treated with PBSO who choose HRT have a comparable overall survival and specific survival for breast / gynecological cancer to women who undergo surgery and refuse to receive HRT.
3. Premenopausal mutation carriers treated with PBSO have better overall and specific breast / gynecological cancer survival than non-SOBP carriers.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 and 49 years
2. Being a member of a family with a history of hereditary breast and ovarian cancer, with a cancer risk> 10% or being a carrier of the BRCA1 / 2 or PALB2 mutation.

Exclusion Criteria:

1. Personal history of oophorectomy for benign or malignant ovarian pathology.
2. Personal history of breast cancer.

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women identified and followed at the Hospital de la Santa Creu i Sant Pau.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
To compare the scale MenCav of quality of life in premenopausal carriers opting and rejecting hormone replacement therapy post salpingo-oophorectomy | 5 years
  Questionnaire to measure quality of life in post-menopausal women (the Mencav questionnaire). This questionnaire consists of questions with 5 possible answers, answer 1 is the worst result and question 5 is the best result, so low scores mean worse results and high scores better results.

SECONDARY OUTCOMES:
To compare the impact of hormone replacement therapy on number and description of cardiovascular events | 5 years
  To describe cardiovascular risk we used changes in the weight of patients. Weight in kilograms, height in meters and weight and height will be combined to report BMI in kg/m^2.
To compare the impact of hormone replacement therapy on number and description of cardiovascular events | 5 years
  To describe cardiovascular risk we used changes in blood pressure (mmHg)
To compare the impact of hormone replacement therapy on number and description of cardiovascular events | 5 years
  To describe cardiovascular risk we used changes in lipids levels (cholesterol, triglycerides, HDL, LDL and VLDL)
To compare the impact of hormone replacement therapy on number and description of cardiovascular events | 5 years
  To describe cardiovascular risk we used eventual cardiovascular adverse events
To compare the impact of hormone replacement therapy on number and description of bone loss related events in premenopausal carriers after salpingo-oophorectomy we will perform bone densitometry | 5 years
  By performing bone densitometry we will be able to quantify the number of participants with adverse events related to bone loss (osteoporosis or osteopenia)
Comparison of overall cancer survival between women deciding risk-reducing surgery and those rejecting it. | 5 years
  We will analyze and compare the mean of overall survival of women undergoing for risk-reducing surgery and those rejecting it
Comparison of mean of breast cancer specific survival between women deciding gynecological surgery and those rejecting surgery. | 5 years
  We will analyze and compare the mean of breast cancer specific survival in women undergoing surgery and those rejecting it.
Comparison of gynecologic cancer survival between women deciding preventive surgery and those rejecting it. | 5 years
  We will analyze and compare the mean of gynecologic cancer survival of women undergoing surgery and those rejecting it.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ramon y Cajal, MD PhD, Principal Investigator — Hospital Santa Cruz y San Pablo
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain